CLINICAL TRIAL: NCT04307238
Title: Infrared Pupillometry - Effects of Different Types of General Anesthesia on Postoperative Pupillary Reactivity
Brief Title: Effects of Different Types of General Anesthesia on Postoperative Pupillary Reactivity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Marita Windpassinger M.D., Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1520/2019
Record Dates: First submitted 2019-11-22; First posted 2020-03-13 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Pupillary Reflex Impaired
Keywords: Pupillary Light Reflex; General Anesthesia; Postoperative Vigilance; Alertness; Postoperative Recovery; Infrared Pupillometry

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blinded study design (participants, evaluator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol group (Other): General anesthesia will be maintained by continually intravenous administered propofol.
  Interventions: Diagnostic Test: PLR; Diagnostic Test: Alertness testing; Procedure: Propofol anesthesia
- Sevoflurane Group (Other): General anesthesia will be maintained by inhalative administered sevoflurane.
  Interventions: Diagnostic Test: PLR; Diagnostic Test: Alertness testing; Procedure: Sevoflurane anesthesia

INTERVENTIONS:
Diagnostic Test: PLR — PLR measurements will be performed within the first 2 postoperative hours.
  Other Names: Pupillary light reflex
Diagnostic Test: Alertness testing — Preoperative (baseline) and every 30 minutes postoperative computer based alertness testing will be performed.
  Other Names: DSST, VIA, TMT
Procedure: Propofol anesthesia — Maintenance of anesthesia will be performed using propofol.
  Arms: Propofol group
Procedure: Sevoflurane anesthesia — Maintenance of anesthesia will be performed using sevoflurane.
  Arms: Sevoflurane Group

SUMMARY:
Objective: To compare the effects of volatile and intravenous anesthetics on pupillary function after general anesthesia using a portable infrared pupillometer.

Design: A monocentric, prospective, double blinded randomized study.

Patients: Patients who require elective Ear, Nose and Throat (ENT) surgery under general anesthesia.

Interventions: Patients undergoing elective ENT surgery will be assigned to intravenous versus inhalative anesthesia and pupillometric parameters monitored postoperative, using an infrared pupillometer.

Outcomes measures: Reported pupillometric parameters after intravenous and inhalative anesthesia.

The purpose of this study is to compare general anesthesia techniques (volatile, intravenous) on postoperative changes in pupillary reactivity by using infrared pupillometry.

DETAILED DESCRIPTION:
Introduction: With the increased focus on early discharge after surgery and anesthesia, it is important to identify objective criteria that can be used to assess home-readiness after ambulatory surgery. Premature discharge may lead to a higher rate of patients suffering complications and to an increased readmission rate. Time-consuming objective evaluations of postoperative vigilance status like EEG registrations are not practicable in routine postoperative clinical practice.

In this study an approach to a more quantitative judgment of postoperative vigilance and consciousness is made by recording pupillometric measurements using a portable infrared pupillometer. The findings of this study may provide new important insights to the meaning of pupillary responses for postoperative vigilance measurement.

Aim: With regard to the lack of knowledge about mechanisms that enable the central nervous system to restore consciousness after the deep functional disorder of the anesthetized state, this study aims to compare general anesthesia techniques (volatile, intravenous) on postoperative changes in pupillary reactivity by using infrared pupillometry.

The primary aim of this study is to investigate changes in pupillary reactivity (pupillary light reflex (PLR, %) in the early postoperative phase (2 hours) after common used types of general anesthesia techniques (inhaled - sevoflurane versus intravenous - propofol).

Secondary aim is to examine whether decreased postoperative PLR predicts a decline in neuropsychological testing (alertness).

Hypotheses: The investigators hypothesis that changes in PLR within the first 2 postoperative hours differs depending on the anesthesia technique used, with a lower decline in PLR after propofol compared to sevoflurane anesthesia.

Furthermore, the investigators hypothesis that postoperative PLR correlates with changes in alertness measured by a neuropsychological test.

Design: This study will be a prospective, randomized double blinded study.

Methods: The study is approved by the local ethics committee and written informed consent will be obtained from each patient. A total of 108 patients aged ≥18 and ≤99 years, with American Society of Anesthesiologist (ASA) physical status scores I-II, scheduled for elective ENT surgery will be enrolled. Baseline assessment of pupillometry and neuropsychological test will be carried out before surgery (baseline) and at predefined time intervals during the first 2 postoperative hours after the end of anesthesia. Results (AUC, PLR%) will be compared between both anesthesia groups.

Primary outcome parameter will be the AUC of PLR (percentage change, %) measured every 15 minutes during the first 2 postoperative hours. Secondary outcome parameter will include the neuropsychological test score (Digit Symbol Substitution Test (DSST), the Visual Intrinsic Alertness Test (VIA) and the Trail making Test (TMT)) will be performed every 30 minutes after general anesthesia (sevoflurane, propofol maintained).), assessed every 30 min up to 2 hours after discontinuation of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 and ≤99 years
* ASA I-II
* Patients undergoing elective ENT surgery under general anesthesia

Exclusion Criteria:

* Patients aged < 18 and >99 years
* consumption of antidepressants, tranquilizer, psychotropic medications
* history of mental illness, neurosurgery, neurological or psychiatric disease
* ophthalmologic disease
* preexisting cognitive impairment
* Patients with drug dependence, alcoholism
* the patients' inability to follow procedures
* implanted electronic medical devices

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2020-03-09 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
The AUC of Pupillary Light Reflex | baseline and within the first 2 postoperative hours
  The AUC of PLR (percentage change, %) measured every 15 minutes during the first 2 postoperative hours.

SECONDARY OUTCOMES:
Alertness assessed with the Visual Intrinsic Alertness Test Score | baseline and within the first 2 postoperative hours
  Neuropsychological test scores of the Visual Intrinsic Alertness Test (VIA) will be assessed every 30 min up to 2 hours after general anesthesia (sevoflurane, propofol maintained).During the VIA test, the participant has to press a button as fast as possible whenever a black circle (diameter 30 mm) appears in the centre of the computer screen. The circle appears for 1500 ms and disappears if no response is given within this time interval. Interstimulus intervals vary between 3-5 s. The tests used are standardised and scores are measured in milliseconds, higher values/scores mean a worse outcome.
Alertness assessed with the Trail making Test Score | baseline and within the first 2 postoperative hours
  Neuropsychological test scores of the Trail making Test (TMT) will be assessed every 30 min up to 2 hours after general anesthesia (sevoflurane, propofol maintained). The TMT test consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible. In the first part, the targets are all numbers (1, 2, 3, etc.) and the test taker needs to connect them in sequential order. In the second part, the subject alternates between numbers and letters (1, A, 2, B, etc.). If the subject makes an error, the test administrator corrects them before the subject moves on to the next dot.
  The goal of the test is for the subject to finish both parts as quickly as possible, with the time taken to complete the test being used as the primary performance metric. The tests used are standardised and scores are measured in seconds, higher values/scores mean a worse outcome.
Alertness assessed with the Digit Symbol Substitution Test | baseline and within the first 2 postoperative hours
  Neuropsychological test scores of the Digit Symbol Substitution Test (DSST) will be assessed every 30 min up to 2 hours after general anesthesia (sevoflurane, propofol maintained). Scores range from 0 to 100, with higher scores indicating higher cognitive function.
  The DSST test consists of 9 digit-symbol pairs (e.g. 1/-,2/┴ ... 7/Λ,8/X,9/=) followed by a list of digits. Under each digit the subject should write down the corresponding symbol as fast as possible. The number of correct symbols within the allowed time (90 sec) is measured. The tests used are standardised and scores are measured in seconds, higher values/scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Vienna, Austria